CLINICAL TRIAL: NCT04300634
Title: Encouraging Physical Activity: Action Or Direction?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eren Avcıl, Physiotherapist, MSc, Istanbul University - Cerrahpasa
Other Study IDs: 001
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Healthy Children and Their Parents
Keywords: physical activity; active children; active parents
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children whose parents are physiotherapists: The demographic data of the child and the parent whom he/she played a role in will be recorded. The physical activity habits of the child and the parent, the sports areas he/she is interested in and the level of activity will be questioned. Physical Activity Questionnaire for Older Children (PAQ-C) and the Physical Activity Diary will be used to assess children's physical activity level. Parameters such as physical activity status, participation in a regular sports activity, daily average time spent with activity at school and during breaks, daily time allocated to the activity will be evaluated. The International Physical Activity Questionnaire (IPAQ) and Physical Activity Diary will be used to evaluate the level of physical activity of the parents.
- Children whose parents are athletes: The demographic data of the child and the parent whom he/she played a role in will be recorded. The physical activity habits of the child and the parent, the sports areas he/she is interested in and the level of activity will be questioned. Physical Activity Questionnaire for Older Children (PAQ-C) and the Physical Activity Diary will be used to assess children's physical activity level. Parameters such as physical activity status, participation in a regular sports activity, daily average time spent with activity at school and during breaks, daily time allocated to the activity will be evaluated. The International Physical Activity Questionnaire (IPAQ) and Physical Activity Diary will be used to evaluate the level of physical activity of the parents.
- Parents of children who are atletes: The demographic data of the child and the parent whom he/she played a role in will be recorded. The physical activity habits of the child and the parent, the sports areas he/she is interested in and the level of activity will be questioned. Physical Activity Questionnaire for Older Children (PAQ-C) and the Physical Activity Diary will be used to assess children's physical activity level. Parameters such as physical activity status, participation in a regular sports activity, daily average time spent with activity at school and during breaks, daily time allocated to the activity will be evaluated. The International Physical Activity Questionnaire (IPAQ) and Physical Activity Diary will be used to evaluate the level of physical activity of the parents.
- Parents of children who are physiotherapist: The demographic data of the child and the parent whom he/she played a role in will be recorded. The physical activity habits of the child and the parent, the sports areas he/she is interested in and the level of activity will be questioned. Physical Activity Questionnaire for Older Children (PAQ-C) and the Physical Activity Diary will be used to assess children's physical activity level. Parameters such as physical activity status, participation in a regular sports activity, daily average time spent with activity at school and during breaks, daily time allocated to the activity will be evaluated. The International Physical Activity Questionnaire (IPAQ) and Physical Activity Diary will be used to evaluate the level of physical activity of the parents.

SUMMARY:
Children's physical activity level is decreasing globally. Habits acquired in childhood and adolescence tend to continue in adulthood. Therefore, to obtain individuals who do physical activity or sports, this habit should be gained in childhood.

It is necessary to understand the factors affecting children's lives to increase the physical activity level of the children and make the active lifestyle a habit. These factors can be divided into the environment and family. It is the place where the family socialization process begins first and social norms and cultural values are learned. Parents can be more effective than the environment because they are the main decision-makers on the child. Parents configure the child's time, duties, provide the sports equipment to their child, transfer them for activity. They can support an active lifestyle by taking role models by children. Role modeling is defined as the child's behaviors of observation and social learning and their parents' behavior. In a review, it has been reported that physically active parents encourage their children to have more activities and may have active children. Small-group studies using an objective method are limited in terms of generalizability. While determining the activity level of the child and the family, the fact that the families can respond biased for their children and that the mother or father can take a role model according to the gender of the child reduces the quality of the studies. It remains unclear how and to what extent parents affect children's activity levels.

The aim of this study is to compare the physical activity level of children between 9-14 years of age, who have similar physical activity awareness, athletes and physiotherapist parents

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 9-14
* Being literate in Turkish
* Not having any physical disability preventing them from doing physical activities
* Attending physical education class regularly

Exclusion Criteria:

* Having a serious cognitive impairment
* Going to school on foot
* Physiotherapists to be selected for the physiotherapist group to work in the field of sports

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 9-14 years of age, who have similar physical activity awareness, athletes and physiotherapist parents.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-16 (Estimated); Primary Completion 2020-05-16 (Estimated); Study Completion 2020-06-16 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Questionnaire for Older Children (PAQ-C) | 4 weeks
  Physical Activity Questionnaire for Older Children, developed in 2004 by Kowalski et al., is one of the frequently used scales for evaluating children's physical activities. The survey consists of 10 items and the first 9 items are used to calculate activity scores. The 10th item evaluates whether the child participated in the activity in the previous week, depending on the disease or other condition. While the minimum total score is 9, the maximum score is 45. The higher scores indicate that there is more physical activity and the lower scores indicate less physical activity.
Physical Activity Diary | 4 weeks
  A physical activity diary is frequently used in Turkish validity and reliability studies of physical activity surveys. In our study, Physical Activity Diary will be used for children and parents. The activities of the children will be evaluated in the morning, noon and evening for each day for 1 week. The children are asked to fill in the 'sitting, walking, running, jumping, doing sports and being active' activities for each of the morning, lunch and evening slices. It should be noted that the diary can be filled in hours or minutes. Parents' seating, walking, and sports activities are questioned weekly, within and outside the workplace.

SECONDARY OUTCOMES:
The International Physical Activity Questionnaire (IPAQ) | 4 weeks
  The International Physical Activity Questionnaire (IPAQ) was developed to provide a common tool that can be used to obtain internationally comparable data in determining health-related physical activity. The questionnaire, whose short form is widely used, consists of 4 parts. According to IPAQ, individuals spend "8.0 MET" in "severe physical activities", "4.0 MET in moderate physical activities, and 3.3 MET in" walking ". Scoring is done by multiplying the number of minutes and days of activity with the respective MET values. The total MET value is obtained by adding the scores of the subtitles. The total value is called physical activity value. According to the total score, less than 600 weekly MET values are evaluated as low-level physical activity, between 601-3.000 MET are medium level and more than 3,000 MET are high-level physical activity.